CLINICAL TRIAL: NCT03640910
Title: A Cluster-randomized Multicenter Trial Comparing OT-Equator® Versus Locator® Attachments to Retain an Early Loaded Implant Overdenture on Two or Three Implants
Brief Title: Attachment Systems for Implant Overdenture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Rhein 83 Srl (Industry)
Responsible Party: Principal Investigator, Marco Tallarico, Principal advisor, Rhein 83 Srl
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: In_Vitro_Eq_Loc_Smart
Record Dates: First submitted 2018-03-29; First posted 2018-08-21 (Actual); Last update posted 2021-02-09 (Actual); Status verified 2021-02

CONDITIONS: Dental Implants; Dental Prosthesis Failure
Keywords: Dental implants; Overdenture; Randomized controlled trial

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- OT Equators® (Rhein83) (Experimental): After gingival healing the newest low-profile OT Equators® (Rhein83) will be screwed on to the implants, using the OT Equator® square screwdriver (Rhein83), with a torque range of 22-25 N cm. The cuff heights ranged from 0.5 to 7.0 mm, depending on the height of the transition zone of each implant, easily measured using the color-coded millimeter Cuff Height Measurer Gauge (Rhein83) after healing abutment removal.
  Interventions: Device: OT Equators® (Rhein83)
- Locator® (Zest) (Active Comparator): The low-profile attachments Locator® (Zest) will be screwed on to the implants, using the Locator® screwdriver (Zest), with a torque range of 20-25 N cm. The cuff heights of 2.5 or 4.0 mm, depending on the height of the transition zone of each implant, measured using the deep probe of the implant line after healing abutment removal.
  Interventions: Device: Locator® (Zest)

INTERVENTIONS:
Device: OT Equators® (Rhein83) — Attachment systems to retain an implant overdenture
  Arms: OT Equators® (Rhein83)
Device: Locator® (Zest) — Attachment systems to retain an implant overdenture
  Arms: Locator® (Zest)

SUMMARY:
The aim of this randomized controlled trial is to compare peri-implant tissue health, number of complications, and patient's preference between two unsplinted overdenture attachments.

DETAILED DESCRIPTION:
Study design: A cluster-randomized multicenter trial of parallel group design and two arms. Patients with complete edentulous mandible in needed of an implant retained overdenture, will be randomly clustered to receive two or three unsplinted implants. Afterwards, patients that have been randomized to receive two implants will be randomized to receive OT Equator® attachment (Rhein'83, Bologna, Italy) in the test group, or Locator® attachment (Zest Anchors LLC, Espandido, CA, USA) in the control group.

Patients will be selected and consecutively treated in 10 private and public (University) centers in Europe, between December 2017 and December 2018. This study will be conducted in accordance with the principles outlined in the Helsinki Declaration of 1964 for biomedical research involving human subjects, as amended in 2013, and will receive ethical approval by Ethical Committees of the various centers. Patients will be duly informed about the nature of the study. A written informed consent form for surgical and prosthetic procedures, as well as for the use of the clinical and radiological data, will be obtained for each patient. The present research will be registered in the Clinical trial.gov and the manuscript will be written according to the CONSORT guidelines.

Any healthy individual (ASA 1 and 2), aged 18 years or older at the time of enrollment, with complete edentulous mandible, or a failing dentition in the mandible, scheduled to receive an implant supported overdenture, will be considered eligible for the study. Exclusion criteria are the general contraindications to oral surgery, pregnancy or nursing, intravenous bisphosphonate therapy, alcohol or drug abuse, heavy smoking (≥ 20 cigarettes/day), radiation therapy to the head or neck region within the last five years, parafunctional activity, untreated periodontitis, and allergy or adverse reactions to the restorative materials.

Preoperative photographs, panoramic x-rays, and periodontal screening have to be obtained for initial screening and evaluation. Hopeless teeth (in the mandible) have to be extracted 3 months before implant placement and new prosthesis delivery. All of the patients will receive a temporary complete removable denture before implant placement, according to the respective functional and esthetic requirements. If the actual complete removable denture is judged accurate from both patients and clinician, it could be used as temporary solution.

On the day of the surgery, a single dose of an antibiotic (either 2 g of amoxicillin or 600 mg of clindamycin or 500 mg of azitromicin or claritromicin if allergic to penicillin) will be administered 1 h before implant placement (2017 AHA). Immediately before surgery, the participants will rinse with a 0.2% chlorhexidine mouthwash for 1 min. Local anesthesia preferred by the surgeon will be administered. Flapless, or a minimally invasive mucoperiosteal flaps will be elevated. Then, the patients will be randomly clustered to receive two or three unsplinted implants according to congealed indication contained in a close enveloped and derived from a pre-generated list. Afterwards, only the patients that will be randomized to receive two implants will be randomized to receive OT Equator® attachment (Rhein'83, Bologna, Italy) in the test group, or Locator® attachment (Zest Anchors LLC, Espandido, CA, USA) in the control group.

Implants have to be placed in the interforaminal region of the mandible according to a one-stage approach.

Three-IRO: center implant will be placed in the midline, and the distal implants were placed 11 mm distal, aligned at a 0-20-degree inclination corresponding to the center implants (with up to an extensive 40 degrees of divergence between implants them).

Two-IRO: implants will be placed in the canine region of the mandible with an interconnecting line approaching parallelism with the terminal mandibular hinge axis, and an extensive 40 degrees of divergence between implants them.

Any brand of implants that provide either Locator® or OT-Equator® abutments can be placed according to the manufacturer suggestions, in order to achieve an insertion torque of at least 35 N cm. The implant lengths will be dictated by the preoperative radiographs. Jaw bone quality will be rated during the dental implant surgery, by the tactile resistance during drilling, allowing an objective evaluation according to the Lekholm & Zarb index.

After surgery, the patients will be instructed to avoid brushing and trauma at the surgical site. A post-surgical cold and soft diet will be recommended. Smokers will be recommended to avoid smoking for 2 weeks days postoperatively, and oral hygiene instructions will be given (Chlorhexidine 0,12% rinses 3 times/day) . Analgesics (600 mg of ibuprofen or other) will be prescribed as needed. Sutures (if present) will be removed after ten days.

The prosthetic procedures will begin eight weeks after implant placement. A reliable, fully extended impressions of both jaws will be taken. Then, a definitive polysulfide-based or polyether impression will be made by using a customized acrylic resin tray, and master cast will be poured with low expansion, class IV gypsum. Intermaxillary relation using registration plates or clinical bite index, functional occlusal analysis, face-bow, and occlusal vertical dimension have to be taken. Master cast and antagonists will be mounted in a semi adjustable articulator and a diagnostic prosthetic setup will be made and tried in the patient's mouth, in which the functional and aesthetic parameters will be evaluated.

A new metal reinforced, complete removable denture will be delivered in both groups within 4 weeks after second surgery, according to an early loading protocol. The healing abutments will be unscrewed and the implant connections have to be disinfected. Randomized attachment system will be placed and tightened according to the manufacturer.

Test Group (OT Equator®)

After gingival healing the newest low-profile OT Equators® (Rhein83) will be screwed on to the implants, using the OT Equator® square screwdriver (Rhein83), with a torque range of 22-25 N cm. The cuff heights ranged from 0.5 to 7.0 mm, depending on the height of the transition zone of each implant, easily measured using the color-coded millimeter Cuff Height Measurer Gauge (Rhein83) after healing abutment removal. Afterward, spaces to accept the female housing steel cage will be prepared in the fitting surface of the removable complete mandibular denture. Silicone protective discs (Rhein83) will be placed over the OT Equator® attachments. Extra-soft (yellow, 600 g) retentive caps will be initially placed in to the female steel housing, attached to the OT Equator and finally fixed to the denture using self-cured acrylic resin while the patient held the dentures in occlusion, directly chairside. After complete polymerization, the denture will be picked up and silicone discs removed. Acrylic excess will be trimmed and the denture will be refined and polished. One month after prosthesis delivery, the yellow retentive caps will be replaced with a stronger type (pink, 1200 g).

Control Group (Locators) The low-profile attachments Locator® (Zest) will be screwed on to the implants, using the Locator® screwdriver (Zest), with a torque range of 20-25 N cm. The cuff heights of 2.5 or 4.0 mm, depending on the height of the transition zone of each implant, measured using the deep probe of the implant line after healing abutment removal. Afterward, spaces to accept the female housing steel cage will be prepared in the fitting surface of the removable complete mandibular denture. Silicone protective white rings (Zest) will be placed over the Locator attachments. Passive black caps will be used to load the attachment. Attached to the Locator and finally fixed to the denture using self-cured acrylic resin while the patient held the dentures in occlusion, directly chairside. After complete polymerization, the denture will be picked up and white rings removed. Acrylic excess will be trimmed and the denture will be refined and polished. Black caps will be removed and blue ones (6N) will be mounted in the steel housing. One month after prosthesis delivery, the retentive caps will be replaced with a pink matrix (12N).

In both groups, the occlusion will be developed to deliver a lingualized occlusion with balanced contacts during function, avoiding any premature contacts. Nevertheless, when the opposing arch is a removable complete denture, the over-jet has to be left purposely broad, from 2 to 5 mm in order to avoid interferences during function. Instructions will be given to the patients, and recall visits will be scheduled for occlusal adjustments and oral hygiene quality control every six months and, for retentive cap replacement, every year.

Outcomes: implant and prosthetic success and survival rate; biologic and technical complications; marginal bone loss; patients' satisfaction (Oral Health Impact Profile, OHIP-22).

ELIGIBILITY:
Inclusion Criteria:

* Any healthy individual (ASA 1 and 2)( (Dexter and Thompson, 2001), aged 18 years or older at the time of enrollment, with complete edentulous mandible, or a failing dentition in the mandible, scheduled to receive an implant supported overdenture, will be considered eligible for the study.

Exclusion Criteria:

* General contraindications to oral surgery, pregnancy or nursing, intravenous bisphosphonate therapy, alcohol or drug abuse, heavy smoking (≥ 20 cigarettes/day), radiation therapy to the head or neck region within the last five years, parafunctional activity, untreated periodontitis, and allergy or adverse reactions to the restorative materials.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-01-01 (Actual); Primary Completion 2020-01-30 (Actual); Study Completion 2020-12-31 (Actual)

PRIMARY OUTCOMES:
Implant and prosthetic success rate | Up to 5 years after implant placement
  An implant will be considered a failure if it presented with any mobility, assessed by tapping or rocking the implant head with the metallic handles of two instruments, progressive marginal bone loss or infection, and any mechanical complications rendering the implant unusable, although still mechanically stable in the bone.

SECONDARY OUTCOMES:
Marginal bone loss | Up to 5 years after implant placement
  Marginal bone levels will be assessed using intraoral digital or conventional periapical radiographs taken with the paralleling technique by means of Rinn-type collimator at implant placement, loading (baseline) and one year after loading. The marginal bone levels will be determined from linear measurements performed by two independent (semi-blinded) trained examiners on each periapical radiograph, from the mesial and distal margin of the implant neck to the most coronal point where the bone appeared to be in contact with the implant.
Oral Health Impact Profile | Up to 5 years after implant placement
  Oral Health Impact Profile(OHIP-19) questionnaire, which will be completed by the participants every year after prosthesis delivery. The questionnaire consists of seven subscales FL = Functional limitation, P1 = Physical pain, P2 = Psychological discomfort, D1 = Physical disability, D2 = Psychological disability, D3 = Social disability, H = Handicap, with two to three questions each. Participants chose from five possible responses for each question as follows: 4= very often; 3= fairly often; 2= occasionally; 1= hardly ever; 0= never/don't know. Lower OHIP total scores are suggestive of improvement in oral health-related quality of life. The questionnaire will be administered before treatment and one month and one year after definitive prosthesis delivery by a blinded examiner.

CONTACTS AND LOCATIONS:
Overall Officials: Marco Tallarico, Dr, Principal Investigator — University of Aldent, Tirana
Locations (1):
- Studio Dr. Marco Tallarico, Rome, Italy